CLINICAL TRIAL: NCT04597008
Title: Topical Antibiotic Therapy to Reduce Infection After Operative Treatment of Fractures at High Risk of Infection: TOBRA - A Multicenter Randomized Controlled Trial
Brief Title: Topical Antibiotic Therapy to Reduce Infection After Operative Treatment of Fractures at High Risk of Infection: TOBRA
Acronym: TOBRA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-19-1-0848
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Post Operative Surgical Site Infection
Keywords: Surgical site infection risk prevention; Bacterial species type and antibacterial sensitivities
MeSH Terms: interventions — Therapeutics; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Standard of Care + Local Vancomycin: Participants in the control group will receive a dose of 1000mg of Vancomycin powder in their wound bed, which is placed right before wound closure at the final stage of definitive fracture fixation.
  Interventions: Drug: Control group
- Treatment (Experimental): Standard of Care + Local Vancomycin + Local Tobramycin: Participants in the treatment group will receive a dose of 1000mg of Vancomycin powder AND a dose of 1200mg of Tobramycin powder in their wound bed, which is placed right before wound closure at the final stafe of definitive fracture fixation.
  Interventions: Drug: Treatment group

INTERVENTIONS:
Drug: Treatment group — Standard of Care + Local Vancomycin + Local Tobramycin: Participants in the treatment group will receive a dose of 1000mg of Vancomycin powder AND a dose of 1200mg of Tobramycin powder in their wound bed, which is placed right before wound closure at the final stafe of definitive fracture fixation.
  Other Names: Treatment
  Arms: Treatment
Drug: Control group — Standard of Care + Local Vancomycin: Participants in the control group will receive a dose of 1000mg of Vancomycin powder in their wound bed, which is placed right before wound closure at the final stage of definitive fracture fixation.
  Other Names: Control
  Arms: Control

SUMMARY:
The overall objective is to compare the effect of Vancomycin and Tobramycin powder combined (treatment) to Vancomycin powder (control) in the reduction of post-fixation infections of tibial plateau and tibial pilon fractures at high risk of infection (collectively considered the "study injuries").

DETAILED DESCRIPTION:
Specific Aim 1: Compare the proportion of deep surgical site infections (SSI) of the study injury within 182 days of definitive fracture fixation surgery in patients allocated to receive a combination of local Vancomycin and Tobramycin powders compared to patients allocated to local Vancomycin powder.

Sensitivity Analyses: A series of sensitivity analyses will be conducted to look at alternative measures of deep SSI under Specific Aim 1. These sensitivity analyses will consider the following alternative end points of deep SSI: infection by only gram-negative bacteria, infection by any gram-positive bacteria (with or without other organisms of any type), polymicrobial pathogenic infections, culture negative infections, and cellulitis/skin infections.

Specific Aim 2: To compare the safety of treatment with a combination of local Vancomycin and Tobramycin versus Vancomycin powder alone as measured by the proportion of antibiotic resistance in each arm.

ELIGIBILITY:
Inclusion Criteria:

1. Tibial plateau or tibial pilon fractures that is treated operatively with plate and screw fixation AND at least one of the following characteristics indicative of higher risk of infection:

   1. Initially treated with an external fixation and treated definitively more than 3 days later after swelling has resolved.
   2. Any open type I, II, or IIIA fracture, regardless of timing of definitive treatment.
   3. Tibia fracture is associated with ipsilateral leg compartment syndrome and fasciotomy wounds.
2. Patients ages 18 through 80 years.

Exclusion Criteria:

1. Study injury is already infected at time of study enrollment.
2. Definitive fixation of the study injury prior to enrollment in the study.
3. The patient never receives study fixation.
4. Massive myonecrosis from ipsilateral leg compartment syndrome.
5. Currently pregnant.
6. Severe problems with maintaining follow-up (e.g. patients who are homeless at the time of injury, those who are intellectually challenged without adequate family support, or are unwilling to provide phone and address contact information).
7. Patients with allergies, drug administration reactions, or other sensitivities to Vancomycin (such as a history of Redman's Syndrome).
8. Patients with allergies, drug administration reactions, or other sensitivities to Tobramycin or other aminoglycosides.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1550 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Deep Surgical Site Infection (SSI) | within 182 days of definitive fracture fixation surgery
  Compare the proportion of deep SSIs of the study injury within 182 days of definitive fracture fixation surgery in patients treated with local Vancomycin powder compared to those treated with a combination of local Vancomycin and Tobramycin powders. For this study a "deep SSI" is a SSI that is treated with operative debridement. In the current CDC terminology this would include all deep organ space, deep incisional, and superficial infections that are treated with surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Robert V O'Toole, MD, MS, Principal Investigator — University of Maryland, Department of Orthopaedic Trauma; Renan C Castillo, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Anthony R Carlini, MS, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (41):
- United States (41):
  - University of Alabama Heersink School of Medicine, Birmingham, Alabama
  - Keck School of Medicine of USC, Los Angeles, California
  - Stanford University, Redwood City, California
  - _University of California, San Francisco, San Francisco, California
  - Cedars Sinai, West Hollywood, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - St Mary's University/Tenent Health, West Palm Beach, Florida
  - Loyola University Chicago, Chicago, Illinois
  - Indiana University School of Medicine - Methodist Hospital, Indianapolis, Indiana
  - Indiana University/Eskenazi Health, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - LSU Health Sciences, New Orleans, Louisiana
  - University of Maryland Shock Trauma Center, Baltimore, Maryland
  - University of Maryland Shock Trauma/Capitol Regions, Baltimore, Maryland
  - Harvard/Mass General/Brigham Hospitals, Boston, Massachusetts
  - Core Well Health, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Dartmouth Hitchcock, Lebanon, New Hampshire
  - New York Presbyterian/Hospital for Special Surgery, New York, New York
  - Jamaica Hospital Medical Center, Queens, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center/Atrium Health Musculoskeletal Health Institute, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - METROHealth, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Penn State College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Rhode Island Hospital/Brown University, Providence, Rhode Island
  - Medical University of South Carolina -, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
  - UTHealth/McGovern Medical School, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax MEdical Campus, Falls Church, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Schrank GM, O'Hara NN, Lee S, Degani Y, Chung S, Carlini AR, Castillo RC, O'Toole RV. Safety of topical tobramycin powder during operative treatment of fractures. J Antimicrob Chemother. 2025 Sep 3;80(9):2417-2420. doi: 10.1093/jac/dkaf230. PMID 40667718